CLINICAL TRIAL: NCT01338116
Title: Optimal Antibiotic Treatment of Moderate to Severe Bacterial Infections: Integration of PCR Technology and Medical Informatics/Artificial Intelligence
Brief Title: Optimal Antibiotic Treatment of Moderate to Severe Bacterial Infections
Acronym: CDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, leibovici leonard, Professor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6036
Record Dates: First submitted 2011-03-30; First posted 2011-04-19 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Community-associated Infections; Health-care Acquired Infections; Nosocomial Infections
Keywords: computerized decision support system; PCR; antibiotic treatment
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Management by TREAT/PCR (Experimental): The data available at the time of patient recruitment will be entered into TREAT. TREAT will provide advice for the empirical antibiotic treatment and unless the caring physician can justify a deviation from this recommendation, TREAT's recommendation will be implemented (yes or no antibiotic treatment and type of antibiotic). TREAT will also recommend whether a blood sample for PCR should be obtained. Blood will be collected aseptically and the test will be performed once daily between 1000AM-1700PM (results available daily at 1700 PM). PCR results and a PCR-revised TREAT recommendation will be reported to the patient's physician in charge and treatment will be revised accordingly.
  Interventions: Other: antibiotic treatment of by TREAT/PCR
- Usual management (No Intervention): Patients will be managed by physicians as in regular clinical practice.

INTERVENTIONS:
Other: antibiotic treatment of by TREAT/PCR — Management by TREAT/PCR. The data available at the time of patient recruitment will be entered into TREAT. TREAT will provide advice for the empirical antibiotic treatment and unless the caring physician can justify a deviation from this recommendation, TREAT's recommendation will be implemented (yes or no antibiotic treatment and type of antibiotic). TREAT will also recommend whether a blood sample for PCR should be obtained. Blood will be collected aseptically and the test will be performed once daily between 1000AM-1700PM (results available daily at 1700 PM). PCR results and a PCR-revised TREAT recommendation will be reported to the patient's physician in charge and treatment will be revised accordingly. On day 2, when results of blood cultures and other cultures become available TREAT will be re-consulted and will issue a new recommendation based on the full microbiological investigation (negative and positive results).
  Arms: Management by TREAT/PCR

SUMMARY:
Severe bacterial infections are associated with mortality of about 30%. Patients with moderate to severe bacterial infections given early and appropriate empirical antibiotic treatment are at a lesser risk for a fatal outcome, with odds ratios ranging from 1.6 to 6.9. However only about 2/3 of patients worldwide are given early and appropriate empirical antibiotic treatment. About 40% of patients treated with antibiotics are given superfluous treatment.

TREAT is a computerized decision support system for antibiotic treatment in inpatients with common bacterial infections. TREAT is based on a state of the art stochastic model of the domain (a causal probabilistic network) and uses a cost benefit model for antibiotic treatment, including costs assigned to future resistance. It was tested in a randomized controlled trial in 3 countries and shown to improve the percentage of appropriate empirical antibiotic treatment while at the same time reduce hospital stay and the use of broad-spectrum antibiotics. The main limitation of TREAT is inherent in the limited information available within hours of presentation.

A second attractive approach to improve antibiotic treatment is to use techniques that do not depend on cultures, and thus shorten the time to identification of the pathogen to a few hours only. The LightCycler® SeptiFast test from Roche performs in vitro nucleic acid amplification test for pathogens causing bloodstream infections.

The purpose of the clinical trial is to show that the combined system TREAT/PCR assays will improve the outcome of inpatients with moderate to severe bacterial infections, while at the same time reducing the use of broad-spectrum antibiotics, with no or little additional costs. A secondary objective will be to assess the sensitivity and specificity of whole blood PCR, using TREAT as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

The rationale of the study will be to address patients for whom antibiotic treatment is, or should be, considered. Thus we will include consecutive patients detected in medical departments according to the following criteria:

1. Patients from whom blood cultures were drawn or
2. All patients for whom antibiotic treatment (but not prophylaxis or intra-peritoneal, inhalation or local antibiotics therapy ) is started within the last 96 days or
3. Patients fulfilling the CDC diagnostic criteria for any infection (see appendix C) or
4. Patients with temperature ≥38.3 measured orally (or 38 axillary or 38.5 rectal) on a single measurement or ≥38 / < 36 on at least 2 consecutive measurements separated at least 1 hr apart and one of the next criteria:

   (a) heart rate >90 beats/minute; (b) respiratory rate >20 breaths/minute or partial pressure of CO2 <32 mm Hg; and (c) white blood cell count >12,000/ L, <4000 L, or >10% immature (band) forms. or
5. Patients with shock compatible with septic shock. As defined as hypotension (arterial blood pressure <90 mmHg systolic, or 40 mmHg less than patient's normal blood pressure) for at least 1 h despite adequate fluid resuscitation; Or Need for vasopressors to maintain systolic blood pressure >90 mmHg or mean arterial pressure >70 mmHg and a suspected source of infection.

Exclusion Criteria:

1. HIV positive patients with opportunistic infection (suspected or proven)and / or AIDS defining illness in the last 6 months prior to data collection.
2. Children<18 years.
3. Suspected travel infections.
4. Suspected tuberculosis.
5. Pregnancy.
6. We will exclude patients not able to sign informed consent or not having a legal guardian willing to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-04; Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Clinical success defined as 30-day survival and clinical stability on day 4 | 30 days
  patient alive at day 30; on day 4: no fever, no intra-tracheal tube, hemodynamic stable, no vasopressor support, empirical treatment appropriate (and thus not changed).

SECONDARY OUTCOMES:
Appropriate empirical antibiotic treatment | 48 hours
  Appropriateness of the antibiotic treatment given during the first 48 hours, before identification of the causative pathogen and its antibiotic susceptibilities
Survival | 30 days
Hospital stay | 30 days
  Length of hospital stay
Antibiotic miuse of broad spectrum antibiotics and total costs of antibiotic treatment Superfluous antibiotic treatment | 30 days
  Use of broad spectrum antibiotics and total costs of antibiotic treatment
Costs | 30 days
  Costs incurred during hospital stay
Adverse events | 30 days
  Allergy, nephrotoxicity, diarrhea, clostridium-difficile associated diarrhea and others

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rabin Medical Center; Leonard Leibovici, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikvah, Israel